CLINICAL TRIAL: NCT03550079
Title: the Fixation Method for the Treatment of Femoral Neck Fractures
Brief Title: Fixation for the Treatment of Femoral Neck Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11156458
Record Dates: First submitted 2018-04-23; First posted 2018-06-08 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Femoral Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three screws fixation (Experimental): femoral neck fractures were fixed with three converted screws
  Interventions: Procedure: fixation
- four screws fixation (Experimental): femoral neck fractures were fixed with four screws
  Interventions: Procedure: fixation

INTERVENTIONS:
Procedure: fixation — treated with different fixation method

SUMMARY:
The femoral neck fracture is the most prevalent injuries which commonly encountered among older people with high mortality, morbidity and young fit healthy ones who subjected to high-energy trauma . Non-union or avascular necrosis of femoral neck fracture which lead to loss of labor capacity and death, is the most commonly occurred complication and results in considerable burden for family. The treatment is difficult and challenging, and to minimize the negative results such as limited mobilization or other complications, it is essential to take active prevention and appropriate treatment depending on fracture pattern and patients' characteristics as early as possible. However, current implant selections for femoral neck fractures remain a topic of greater interest and controversy, and vary substantially from each other .

DETAILED DESCRIPTION:
The incidence of femoral neck fracture accounts for 3.6% of all fractures, is the most prevalent injuries which commonly encountered among older people with high mortality, morbidity and young fit healthy ones who subjected to high-energy trauma . Non-union or avascular necrosis of femoral neck fracture which lead to loss of labor capacity and death, is the most commonly occurred complication and results in considerable burden for family. The treatment is difficult and challenging, and to minimize the negative results such as limited mobilization or other complications, it is essential to take active prevention and appropriate treatment depending on fracture pattern and patients' characteristics as early as possible. However, current implant selections for femoral neck fractures remain a topic of greater interest and controversy, and vary substantially from each other depending on the extent of displacement, fracture configuration, physiological age of the patient, bone quality or other relative factors. Nonoperative management is considered only when patients are seriously ill or presented with excessive surgical risk.

ELIGIBILITY:
Inclusion Criteria:

* closed femoral neck fracture
* no fractures at other sites
* surgical treatment with cannulated compression screws or PFNA
* follow-up time greater than 1 years.

Exclusion Criteria:

* the absence of severe cognitive dysfunction,
* the presence of a pathological femoral neck fracture
* previous femoral neck fracture, treated with other internal fixations and surgical treatment with open reduction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
outcome measure were evaluated by femoral neck shortening with X rays | up to 12 months
  femoral neck shortening after 1 year with radiology measure,

SECONDARY OUTCOMES:
nonunion | up to 12 months
  the number of nonunion at the end of follow up in patients
screw-exit | up to 12 months
  screw-exit afer 1 year with X rays in all patients
cut-out | up t 12 months
  cut-out of the screw evaluating with x rays in all patients

OTHER OUTCOMES:
operative time in every patient | intraoperation
  outcome measure were evaluated by operative time
fluoroscopy time intraoperatively | intraoperation
  outcome measure were evaluated by operative time and fluroscopy time

CONTACTS AND LOCATIONS:
Overall Officials: zhiyong Hou, MD, Study Director — Hebei Medical University Third Hospital
Locations (1):
- the Third Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
the data should be allowed by Zhang Yingze

REFERENCES:
- [Derived] Guo J, Dong W, Yin B, Jin L, Lin Z, Hou Z, Zhang Y. Intramedullary nails with cannulated screw fixation for the treatment of unstable femoral neck fractures. J Int Med Res. 2019 Feb;47(2):557-568. doi: 10.1177/0300060518816185. Epub 2018 Dec 11. PMID 30526163